CLINICAL TRIAL: NCT01987908
Title: A Phase 2, Exploratory, Placebo-Controlled, Multicenter, Double-Blind Evaluation of the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Effects of Two Dose Regimens of Aes-103 Given for 28 Days to Subjects With Stable Sickle Cell Disease
Brief Title: Evaluation of Different Dose Regimens of Aes-103 Given for 28 Days to Subjects With Stable Sickle Cell Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early by the Sponsor due to unblinding between study drug and placebo groups at the subject, site and Sponsor levels.
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Aes-103-003; 321401 (Other: Baxalta); 2013-001534-18 (EudraCT Number)
Record Dates: First submitted 2013-10-29; First posted 2013-11-20 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Sickle Cell Disease
Keywords: Pain; Biomarkers; 6 minute walk test; 5-HMF; Pharmacokinetics; Analgesic use; Sickle cell disease; Aes-103; SpO2; Anemia; Hemoglobin
MeSH Terms: conditions — Anemia, Sickle Cell; Pain; Anemia | interventions — 5-hydroxymethylfurfural

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort A (Drug) (Experimental): Subjects randomized 3:1 to receive 4 times daily dosing of 1,000 mg of Aes 103 or placebo for 28 days
  Interventions: Drug: Aes-103
- Cohort A (Placebo) (Placebo Comparator): Subjects randomized 3:1 to receive 4 times daily dosing of 1,000 mg of Aes 103 or placebo
  Interventions: Other: Placebo
- Cohort B (Drug) (Experimental): In this adaptive design, the dose frequency and the total amount given per day to Cohort B will be adjusted depending on the tolerability, clinical pharmacology and clinical endpoint results of Cohort A. Study terminated prior to completion of Cohort A due to unblinding between study product and placebo groups for participant, site and Sponsor. The study was stopped before initiation of Cohort B.
  Interventions: Drug: Aes-103
- Cohort B (Placebo) (Placebo Comparator): The dosing regiment of placebo will match that of the Aes-103 treatment in Cohort B. Study terminated prior to completion of Cohort A due to unblinding between study product and placebo groups for participant, site and Sponsor. The study was stopped before initiation of Cohort B.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aes-103 — The active ingredient in Aes-103 is 5-hydroxymethyl furfural (5-HMF). Aes-103 and matching placebo are administered in a liquid oral formulation.
  Arms: Cohort A (Drug); Cohort B (Drug)
Other: Placebo
  Arms: Cohort A (Placebo); Cohort B (Placebo)

SUMMARY:
Sickle cell disease (SCD) is a genetic blood disorder characterized by the presence of sickle-shaped red blood cells. In the U.S. and the U.K. this occurs primarily in persons of African origin. There is only one drug (hydroxyurea) approved to manage SCD, but it is not fully efficacious and can produce medically significant side effects. Aes-103 is being evaluated as a novel agent for the long term management of SCD. By directly reducing the sickling process, Aes-103 has a different mechanism of action than hydoxyurea. The active ingredient in Aes-103 is 5-hydroxymethyl furfural, a naturally occurring small molecule that is chemically related to glucose.

This study will evaluate the safety and pharmacokinetic profile of two dosing regimens of Aes-103 for up to 28 days in up to 50 adult subjects with stable SCD compared with subjects receiving placebo.

DETAILED DESCRIPTION:
This study will evaluate evaluate in subjects with stable SCD the safety, pharmacokinetic profile, clinical pharmacology actions and clinical activities of two dosing regimens of Aes-103 (1000 mg four times daily in Cohort A and a higher or lower dose given once daily or up to four times daily in Cohort B) given for up to 28 days in adult subjects with stable SCD compared with subjects receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-60 years old, inclusive
* Diagnosis of SCD (hemoglobin SS) without hospitalization for pain crises or any other reason in the 14 days before enrollment
* Have normal organ function as defined by direct bilirubin <1.1 mg/dL (19 μmol/L), alanine transaminase (serum glutamic pyruvic transaminase) ≤120 IU/L, and Creatinine ≤1.3 mg/dL (115 μmol/L)
* Have at least one of the following baseline values: hemoglobin level of <10 g/dL, numerical pain rating scale (NPRS) score of ≥ 4, or 6-minute walk distance (6MWD) of <500 m
* If female, be nonpregnant and nonbreastfeeding and be surgically sterile or using an acceptable method of contraception throughout the study and for 3 months after the last dose of study medication
* Have completed an outpatient screening visit consisting of medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs, hematology and chemistry tests, urinalysis, urine drug screen, urine or serum pregnancy test (females), hemoglobin electrophoresis, hepatitis B and C screening, and HIV serology
* Be able to understand and have provided written informed consent including signature on an informed consent form approved by an institutional review board or independent ethics committee
* Have provided written authorization for use and disclosure of protected health information
* Agree to abide by the study schedule and to return for the required assessments

Exclusion Criteria:

* Have been hospitalized in the 14 days before enrollment, for any reason
* Have evidence of clinically significant cardiovascular, respiratory, renal, hepatic, pulmonary, gastrointestinal, hematological, neurological, psychiatric, or other disease that may interfere with the objectives of the study or the safety of the subject, or have been hospitalized in the past 6 months as a result of these conditions (for SCD-related morbidity, a minimum of 14 days from the last hospitalization is required)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2015-03-16 (Actual); Study Completion 2015-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Quintiles Ltd. - Quintiles Drug Research Unit, 6 Newcomen Street, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at one clinical site in the United Kingdom with referrals and/or patient identification from five other clinical sites in the United Kingdom.
Pre-assignment Details: 35 participants were enrolled. 10 failed screen and 2 were randomization failures. 23 started the 2-week, single-blind, placebo lead-in period (to obtain stable baseline values and to screen out participants who did not tolerate placebo or were not compliant with study procedures).
Groups:
- Placebo lead-in Period: Participants enrolled in a 14 day single-blind placebo lead-in received 4 times daily dosing of placebo
- Treatment With Study Product: After placebo lead-in period, participants randomized 3:1 (Aes-103 to placebo) to receive 4 times daily dosing of 1,000 mg of Aes-103 for 28 days during the double-blind treatment period
- Treatment With Placebo: After placebo lead-in period, participants randomized 3:1 (Aes-103 to placebo) to receive 4 times daily dosing of 1,000 mg of placebo for 28 days during the double-blind treatment period
Period: Placebo Lead-in Period
Arm/Group | Placebo lead-in Period | Treatment With Study Product | Treatment With Placebo
Started | 23 | 0 | 0
Completed | 14 | 0 | 0
Not Completed | 9 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Other: Study Termination by Sponsor | 4 | 0 | 0
Period: Treatment Period
Arm/Group | Placebo lead-in Period | Treatment With Study Product | Treatment With Placebo
Started | 0 | 11 | 3
Completed | 0 | 10 | 2
Not Completed | 0 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 1
Period: Post-Treatment Observation Period
Arm/Group | Placebo lead-in Period | Treatment With Study Product | Treatment With Placebo
Started | 0 | 10 | 2
Completed | 0 | 7 | 2
Not Completed | 0 | 3 | 0
Not completed — Other: Study Termination by Sponsor | 0 | 2 | 0
Not completed — Other: Bad Veins | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Out of the participants who enrolled in the study, only participants who passed the screen and were randomized were entered in the Placebo Lead-in Period.
Arm/Group | Placebo lead-in Period
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events, Including Sickle Cell-specific Symptoms, During the Double-blind Treatment Period
Description: Number of participants with adverse events (AEs) reported during the double-blind treatment period. AEs included clinically-significant changes in vital signs, ECG, clinical laboratory assessments, physical and neurological examinations. Sickle cell-specific symptoms included the development of new skin ulcers, hospitalization or ambulatory acute care, intravenous analgesics visit for pain episodes (i.e., sickle-cell disease related pain), acute chest syndrome, priapism, and stroke.
Time Frame: Double-blind treatment period of 28 days (Day 1 to Day 28)
Measure: Number; unit: participants
Groups:
- Treatment With Study Product: Participants randomized 3:1 (Aes-103 to placebo) to receive 4 times daily dosing of 1,000 mg of Aes-103 for 28 days
- Treatment With Placebo: Participants randomized 3:1 (Aes-103 to placebo) to receive 4 times daily dosing of 1,000 mg of placebo for 28 days
- All Treated Participants: All participants randomized 3:1 (Aes-103 to placebo) and received 4 times daily dosing of 1,000 mg AEs-103 or 1,000 mg of placebo for 28 days
Arm/Group | Treatment With Study Product | Treatment With Placebo | All Treated Participants
Number analyzed (Participants) | 11 | 3 | 14
participants
  Treatment-emergent AEs | 9 | 3 | 12
  Related AEs | 8 | 2 | 10
  Serious AEs | 0 | 0 | 0
  Severe AEs | 0 | 0 | 0
  AEs leading to discontinuation | 1 | 1 | 2
  AEs leading to death | 0 | 0 | 0
  Sickle-cell specific complications | 4 | 1 | 5

2. Primary Outcome: Number of Participants With Adverse Events, Including Sickle-cell Specific Symptoms, During the Placebo lead-in Period
Description: Number of participants with adverse events (AEs) reported during the placebo lead-in period. AEs included clinically-significant changes in vital signs, ECG, clinical laboratory assessments, physical and neurological examinations. Sickle cell-specific symptoms included the development of new skin ulcers, hospitalization or ambulatory acute care, intravenous analgesics visit for pain episodes (i.e., sickle-cell disease related pain), acute chest syndrome, priapism, and stroke.
Time Frame: Placebo lead-in period of 14 days (Day -14 to Day -1)
Measure: Number; unit: participants
Arm/Group | Placebo lead-in Period
Number analyzed (Participants) | 23
participants
  Treatment-emergent AEs | 21
  Related AEs | 12
  Serious AEs | 2
  Severe AEs | 2
  AEs leading to discontinuation | 2
  AEs leading to death | 0
  Sickle cell-specific complications | 2

3. Primary Outcome: Number of Participants With Adverse Events, Including Sickle-cell Specific Symptoms, During the Post-treatment Observation Period
Description: Number of participants with adverse events (AEs) reported during the post-treatment observation period. AEs included clinically-significant changes in vital signs, ECG, clinical laboratory assessments, physical and neurological examinations. Sickle cell-specific symptoms included the development of new skin ulcers, hospitalization or ambulatory acute care, intravenous analgesics visit for pain episodes (i.e., sickle-cell disease related pain), acute chest syndrome, priapism, and stroke.
Time Frame: Post-treatment observation period of 21 days (Day 29 to Day 49)
Measure: Number; unit: participants
Groups:
- Post-treatment With Study Product Observation Period: Participants underwent a post-treatment observation period of 21 days during which no study product (Aes-103) was received
- Post-treatment With Placebo Observation Period: Participants underwent a post-treatment observation period of 21 days during which no placebo was received
- All Participants in Post-treatment Observation Period: Participants underwent a post-treatment observation period of 21 days during which no study product (Aes-103) or placebo was received
Arm/Group | Post-treatment With Study Product Observation Period | Post-treatment With Placebo Observation Period | All Participants in Post-treatment Observation Period
Number analyzed (Participants) | 10 | 2 | 12
participants
  Treatment-emergent AEs | 4 | 0 | 4
  Related AEs | 2 | 0 | 2
  Serious AEs | 1 | 0 | 1
  Severe AEs | 1 | 0 | 1
  AEs leading to discontinuation | 0 | 0 | 0
  AEs leading to death | 0 | 0 | 0
  Sickle cell-specific complications | 2 | 0 | 2

4. Primary Outcome: Number of Participants With Sickle-Cell Disease-related Symptoms
Time Frame: Placebo lead-in period of 14 days (Day -14 to Day -1), double-blind treatment period of 28 days (Day 1 to Day 28) and post-treatment observation period of 21 days (Day 29 to Day 49)
Measure: Number; unit: participants
Arm/Group | Placebo Lead-in Period | Treatment With Study Product | Treatment With Placebo | Post-treatment With Study Product Observation Period | Post-treatment With Placebo Observation Period
Number analyzed (Participants) | 23 | 11 | 3 | 10 | 2
participants
  Abdominal Pain - Sickle Pain | 0 | 1 | 0 | 0 | 0
  Exacerbation of Sickle Cell (SC) Disease Pain | 1 | 1 | 0 | 1 | 0
  SC Disease Related Pain | 0 | 3 | 0 | 1 | 0
  SC Pain | 3 | 3 | 1 | 1 | 0
  Intermittent SC Pain | 1 | 0 | 0 | 0 | 0
  SC Crisis | 1 | 0 | 0 | 0 | 0
  Vaso-Occlusive Crisis caused by Chest Infection | 1 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Clinically Significant Observations of Vital Signs, 12-lead ECGs, Clinical Laboratory Assessments, and Physical and Neurological Examinations
Description: Vital signs, 12-lead ECGs, clinical laboratory assessments, and physical and neurological examinations that were deemed clinically significant by the investigator in agreement with the sponsor study director.
Time Frame: Throughout the study period (approximately 9 weeks)
Population: safety analysis dataset
Measure: Number; unit: clinically significant observations
Groups:
- Placebo lead-in Period: Participants enrolled in a 14 day single-blind placebo lead-in received 4 times daily dosing of placebo (Day -14 to Day -1)
- Double-blind Treatment Period - Study Product: Participants randomized 3:1 (Aes-103 to placebo) to receive 4 times daily dosing of 1,000 mg of Aes-103 for 28 days (Day 1 to Day 28)
- Double-blind Treatment Period - Placebo: Participants randomized 3:1 (Aes-103 to placebo) to receive 4 times daily dosing of placebo for 28 days (Day 1 to Day 28)
- Post-treatment Observation Period: Participants underwent a post-treatment observation period of 21 days during which no study product (Aes-103) or placebo was received (Day 29 to Day 49)
Arm/Group | Placebo lead-in Period | Double-blind Treatment Period - Study Product | Double-blind Treatment Period - Placebo | Post-treatment Observation Period
Number analyzed (Participants) | 23 | 11 | 3 | 12
clinically significant observations
  Electrocardiogram T Wave Inversion | 0 | 1 | 0 | 0
  Transaminases Increased | 0 | 0 | 1 | 0

6. Primary Outcome: PK: - Plasma AUC, Cmax, Tmax, and T1/2 of Aes-103 and Its Metabolite, HMFA - RBC Hemolysate AUC (0-8h), Cmax, Tmax, and T1/2 of Aes-103 - Percentage of Hemoglobin Bound to Aes-103
Description: Pharmacokinetic endpoints in the study protocol were as follows:- - Plasma Area under curve (AUC), Maximum plasma concentration (Cmax), time at which Cmax observed (Tmax), and terminal half-life (T1/2) of Aes-103 and its metabolite, 5-hydroxymethyl-2-furoic acid (HMFA) - red blood cell (RBC) hemolysate Area under curve between 0 and 8 hours (AUC [0-8h]), Cmax, Tmax, and T1/2 of Aes-103 - Percentage of hemoglobin bound to Aes-103
Time Frame: PK blood samples were to be taken within 10 minutes before dosing and 0.5, 1, 2, 4, and 6 hours after the first dose of study product on Days 1 and 7 and at the same time points on Day 28 (or early termination)
Population: PK data were not determined as the assay collection method was found to be faulty rendering all samples unevaluable.
Groups:
- Overall Study Arm: Data not collected
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 0

7. Secondary Outcome: Resting Oxygen Saturation as Measured by Oximetry (SpO2) - Change From Baseline
Description: A measure of the amount of oxygen in the blood. Oxygen saturation was determined by pulse oximetry. A pulse oximeter was placed over a nail polish-free finger nail to determine peripheral oxygen saturation (SpO2). Baseline was defined as the most recent value obtained prior to the start of dosing on Day 1 of the double-blind treatment period. A mean change from baseline >0 indicates an increase in oxygen saturation, a mean change <0 indicates a decrease in oxygen saturation. Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: Prior to, during and after the end of dosing in the double-blind treatment period, i.e., at baseline, Day 4, Day 7, Day 14 and Day 28
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
percent saturation
  Day 4 (n=9, 3) | 0 (2) | 4 (5)
  Day 7 (n= 9, 3) | 0 (2) | -4 (8)
  Day 14 (n=8, 2) | 0 (2) | 8 (10)
  Day 28 (n=8, 2) | 0 (3) | 6 (8)

8. Secondary Outcome: Oxygen Binding p50/p20 Value - Change From Baseline
Description: A measure of the ability of hemoglobin to bind oxygen. The p50 is the oxygen level at which 50% of the hemoglobin contains oxygen. The p20 is the oxygen level at which 20% of the hemoglobin contains oxygen. Baseline is defined as the most recent value obtained prior to start of dosing on Day 1 of the double-blind treatment period. Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: During the double-blind treatment period at baseline, Day 1, Day 4 and Day 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
ratio
  Day 1 (n=11, 3) | 0.0 (0.2) | 0.0 (0.2)
  Day 4 (n=11, 3) | 0.0 (0.1) | 0.1 (0.1)
  Day 7 (n=10, 3) | 0.0 (0.2) | 0.0 (0.1)

9. Secondary Outcome: Plasma Erythropoietin (EPO) Levels - Change From Baseline
Description: Erythropoietin (EPO) is a hormone produced by the kidney that promotes the formation of red blood cells by the bone marrow. EPO can be detected and measured in the blood. Baseline defined as the most recent value obtained prior to the start of dosing on Day 1 of the double-blind treatment period. Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: At baseline and Day 28 during the double-blind treatment period
Population: Participants who provided baseline data and at least one other data point for this outcome measure.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
U/L | -5.9 (50.3) | -15.1 (20.4)

10. Secondary Outcome: Hematocrit Levels - Change From Baseline
Description: Baseline defined as the most recent value obtained prior to the start of dosing on Day 1 of the double-blind treatment period. Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: Prior to, during and after the end of dosing in the double-blind treatment period, i.e., at baseline, Day 1, Day 7, Day 14 and Day 28
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
L/L
  Day 1 (n=11, 3) | 0.006 (0.011) | -0.002 (0.007)
  Day 7 (n=9, 3) | 0.007 (0.013) | 0.020 (0.010)
  Day 14 (n=8, 2) | 0.003 (0.013) | -0.006 (0.015)
  Day 28 (n=8, 2) | 0.011 (0.012) | 0.006 (0.007)

11. Secondary Outcome: Lactate Dehydrogenase (LDH) Levels - Change From Baseline
Description: LDH levels were measured as a biomarker for intravascular hemolysis. The results are based on the LDH Total measurement. Baseline defined as the most recent value obtained prior to the start of dosing on Day 1 of the double-blind treatment period. Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: as for outcome 10
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
U/L
  Day 1 (n=11, 3) | 60 (107) | 0 (197)
  Day 7 (n=9, 3) | 71 (101) | -6 (167)
  Day 14 (n=8, 2) | 4 (100) | 689 (1142)
  Day 28 (n=8, 2) | 29 (110) | -69 (91)

12. Secondary Outcome: Hemoglobin Levels - Change From Baseline
Description: A clinical laboratory endpoint that reflects the amount of red blood cells present in the blood. Baseline defined as the most recent value obtained prior to the start of dosing on Day 1 of the double-blind treatment period. Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: Prior to, during and after the end of dosing in the double-blind treatment period, i.e., at baseline, Day 1, Day 4, Day 7, Day 14, Day 21 and Day 28
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
g/L
  Day 1 (n=11, 3) | 0 (5) | -3 (7)
  Day 4 (n=10, 3) | 1 (7) | 3 (3)
  Day 7 (n=10, 3) | -1 (5) | 3 (2)
  Day 14 (n=8, 2) | -2 (5) | -6 (1)
  Day 21 (n=2, 0) | 1 (4) | NA (NA) — Data not collected.
  Day 28 (n=10, 2) | 0 (4) | -2 (5)

13. Secondary Outcome: Reticulocyte Percent- Change From Baseline
Description: Category title includes number of participants with available data (n) for participants treated with study product.
Time Frame: At baseline, Day 1 and Day 7 during the double-blind treatment period
Population: Participants who provided baseline data and at least one other data point for this outcome measure. Summary tables for placebo group not done as data not collected. Study terminated early.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Treatment With Study Product
Number analyzed (Participants) | 2
percent
  Day 1 (n=2) | -0.46 (0.18)
  Day 7 (n=1) | NA (NA) — When number of participants is less than 2, summary statistics are not computed.

14. Secondary Outcome: Direct Bilirubin - Change From Baseline
Description: Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: Prior to, during and after the end of dosing in the double-blind treatment period, i.e., at baseline, Day 1, Day 7, Day 14, Day 21 and Day 28
Measure: Mean (Standard Deviation); unit: mircomoles/L
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
mircomoles/L
  Day 1 (n=11, 3) | 0 (0) | 0 (0)
  Day 4 (n=10, 3) | 0 (0) | 0 (0)
  Day 7 (n=10, 3) | 0 (0) | 0 (0)
  Day 14 (n= 8, 2) | 0 (0) | 0 (0)
  Day 21 (n=2, 0) | 0 (0) | NA (NA) — Data not collected.
  Day 28 (n=10, 2) | 0 (0) | 0 (0)

15. Secondary Outcome: LDH Isoform - Change From Baseline
Time Frame: as for outcome 10
Population: Summary tables for this outcome measure were not done as baseline data missing. Study terminated early.
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: C Reactive Protein Levels - Change From Baseline
Description: Category title includes number of participants with available data (n) for participants treated with study product.
Time Frame: At baseline, Day 1 and Day 7 during the double-blind treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Treatment With Study Product
Number analyzed (Participants) | 2
mg/L
  Day 1 (n=2) | -1.2 (3.0)
  Day 7 (n=1) | NA (NA) — When number of participants is less than 2, summary statistics are not computed.

17. Secondary Outcome: Serum Ferritin Levels - Change From Baseline
Time Frame: At baseline, Day 1 and Day 7 during the double-blind treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mircograms/L
Arm/Group | Treatment With Study Product
Number analyzed (Participants) | 2
mircograms/L
  Day 1 | -4.9 (0.1)
  Day 7 | NA (NA) — When number of participants is less than 2, summary statistics are not computed.

18. Secondary Outcome: N-terminal Pro B-type Natriuretic Peptide (NT-proBNP) Levels- Change From Baseline
Description: Category title includes number of participants with available data (n) for participants treated with study product.
Time Frame: At baseline, Day 1, Day 7, Day 14 and Day 28 during the double-blind treatment period
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Treatment With Study Product
Number analyzed (Participants) | 9
pmol/L
  Day 1 (n=7) | 6 (15)
  Day 7 (n=6) | 6 (97)
  Day 14 (n=6) | 32 (25)
  Day 28 (n=7) | 1 (55)

19. Secondary Outcome: Body Weight - Change From Baseline
Description: A negative change in body weight denotes a weight decrease, a positive change in body weight denotes a weight increase. Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: as for outcome 12
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
kg
  Day 1 (n=11, 3) | -0.2 (0.7) | -0.6 (0.4)
  Day 4 (n=10, 3) | -0.3 (1.6) | -0.4 (0.8)
  Day 7 (n=10, 3) | -0.5 (1.6) | -0.7 (1.3)
  Day 14 (n=8, 2) | 1.1 (0.8) | 0.8 (0.7)
  Day 21 (n=6, 2) | 0.1 (1.4) | 0.5 (0.1)
  Day 28 (n=10, 2) | 0.6 (0.9) | 0.4 (0.4)

20. Secondary Outcome: Exercise Tolerance: 6-Minute Walk Distance During the Double-blind Treatment Period - Change From Baseline
Description: Functional exercise capacity was evaluated by using the 6-minute walk test (6MWT) which measures the distance that a subject can quickly walk on a flat, hard surface in a period of 6 minutes. Guidelines developed by the American Thoracic Society were used for conducting the test and interpreting the results. Baseline defined as the most recent value obtained prior to the start of dosing on Day 1. Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: as for outcome 7
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
meters
  Day 4 (n=9, 3) | -8.5 (38.2) | 20.6 (8.0)
  Day 7 (n=9, 3) | 36.9 (44.6) | 28.3 (24.3)
  Day 14 (n=8, 2) | -0.1 (31.5) | 4.1 (6.1)
  Day 28 (n=8, 2) | -14.9 (41.2) | -8.2 (8.2)

21. Secondary Outcome: Exercise Tolerance: 6-Minute Walk Distance on Day 49 of the Post-treatment Observation Period - Change From Baseline
Description: Functional exercise capacity was evaluated by using the 6-minute walk test (6MWT) which measures the distance that a subject can quickly walk on a flat, hard surface in a period of 6 minutes. Guidelines developed by the American Thoracic Society were used for conducting the test and interpreting the results. Baseline defined as the most recent value obtained prior to the start of dosing on Day 1.
Time Frame: Prior to dosing at baseline and on Day 49 of the post-treatment observation period
Population: Participants who provided baseline data and at least one other data point for this outcome measure.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Post-treatment With Placebo Observation Period: Participants underwent a post-treatment observation period of 21 days during which no study product (placebo) was received
Arm/Group | Post-treatment With Study Product Observation Period | Post-treatment With Placebo Observation Period
Number analyzed (Participants) | 8 | 2
meters | -20.6 (41.3) | -1.1 (3.5)

22. Secondary Outcome: Exercise Tolerance: 6-Minute Walk Distance on Day 49 of the Post-treatment Observation Period - Change From Last Day of Double-blind Treatment Period (Day 28)
Description: Functional exercise capacity was evaluated by using the 6-minute walk test (6MWT) which measures the distance that a subject can quickly walk on a flat, hard surface in a period of 6 minutes. Guidelines developed by the American Thoracic Society were used for conducting the test and interpreting the results.
Time Frame: On last day of double-blind treatment period (Day 28) and on Day 49 of the post-treatment observation period
Population: Participants who provided baseline data and at least one other data point for this outcome measure.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Post-treatment With Study Product Observation Period | Post-treatment With Placebo Observation Period
Number analyzed (Participants) | 8 | 2
meters | -5.6 (63.6) | 7.2 (4.7)

23. Secondary Outcome: Exercise Tolerance: Cardiopulmonary Exercise Test [CPET]
Description: CPET was optional, based on capacity of participant to complete the test.
Time Frame: On last day of double-blind treatment period (Day 28)
Population: Following an external review and report of CPET capabilities of the external service provider, all CPET testing was suspended and the decision made to not collect or analyze CPET data.
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 0

24. Secondary Outcome: Patients´ Global Impression of Change (PGIC) During the Double-blind Treatment Period - Change From Baseline
Description: Participants assessed the change in activity limitations, symptoms, emotions, and overall quality of life by using the 1- to 7-point PGIC scale. The question and scale was as follows: Since beginning treatment at this clinic, how would you describe the change in your sickle cell condition? Please circle the number that matches your overall judgment. -3 - much worse -2 - moderately worse -1 - minimally worse 0 - no change +1 - minimally improved +2 - moderately improved +3 - much improved. Baseline defined as the most recent value obtained prior to the start of dosing on Day 1 of the double-blind treatment period. No values available for placebo group for Day 28. Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: At baseline and once weekly on Days 7, 14, 21, and 28 during the double-blind treatment period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
score on a scale
  Day 7 (n=10, 3) | 0 (1) | 0 (0)
  Day 14 (n=9, 2) | 0 (0) | 0 (0)
  Day 21 (n=8, 2) | 0 (1) | 0 (0)
  Day 28 (n=9, 1) | 0 (1) | NA (NA) — When number of participants is less than 2, summary statistics are not computed.

25. Secondary Outcome: Patients´ Global Impression of Change (PGIC) During the Post-treatment Observation Period - Change From Baseline
Description: Participants assessed the change in activity limitations, symptoms, emotions, and overall quality of life by using the 1- to 7-point PGIC scale. The question and scale was as follows: Since beginning treatment at this clinic, how would you describe the change in your sickle cell condition? Please circle the number that matches your overall judgment. -3 - much worse -2 - moderately worse -1 - minimally worse 0 - no change +1 - minimally improved +2 - moderately improved +3 - much improved. Baseline defined as the most recent value obtained prior to the start of dosing on Day 1 of the double-blind treatment period. Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: At baseline and once weekly on Days 35, 42, and 49 during the post-treatment observation period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post-treatment With Study Product Observation Period | Post-treatment With Placebo Observation Period
Number analyzed (Participants) | 10 | 2
score on a scale
  Day 35 (n=8, 2) | 0 (1) | 0 (0)
  Day 42 (n=10, 2) | 0 (1) | 0 (0)
  Day 49 (n=8, 2) | 0 (1) | 0 (0)

26. Secondary Outcome: Patients´ Global Impression of Change (PGIC) During the Post-treatment Observation Period - Change From Last Day of Double-blind Treatment Period
Description: Participants assessed the change in activity limitations, symptoms, emotions, and overall quality of life by using the 1- to 7-point PGIC scale. The question and scale was as follows: Since beginning treatment at this clinic, how would you describe the change in your sickle cell condition? Please circle the number that matches your overall judgment. -3 - much worse -2 - moderately worse -1 - minimally worse 0 - no change +1 - minimally improved +2 - moderately improved +3 - much improved. Baseline was defined as the most recent value obtained on the last day of the double-blind treatment period. Categories contain Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: At baseline and once weekly on Days 35, 42, and 49 during the post-treatment observation period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post-treatment With Study Product Observation Period | Post-treatment With Placebo Observation Period
Number analyzed (Participants) | 10 | 2
score on a scale
  Day 35 (n=8, 2) | 0 (0) | 0 (0)
  Day 42 (n=10, 2) | 0 (0) | 0 (0)
  Day 49 (n=8, 2) | 0 (0) | 0 (0)

27. Secondary Outcome: Numerical Pain Rating Scale (NPRS): Worst Pain (Weekly Average) in the Double-blind Treatment Period - Change From Baseline
Description: Participants assessed their pain levels by using the 0-10 Numeric Rating Scale: 0 = No pain 1-3 = Mild pain (nagging, annoying, interfering little with activities of daily living [ADLs]) 4-6 = Moderate pain (interferes significantly with ADLs) 7-10 = Severe pain (disabling; unable to perform ADLs A negative mean change denotes a pain decrease. A positive mean change denotes an increase in pain. Baseline was defined as the average of all measures taken from screening through the period prior to start of dosing on Day 1. Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: Participants assessed and recorded their pain level daily. Weekly averages were calculated for the Day 7, Day 14, Day 21, and Day 28 assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
score on a scale
  Day 7 (n=11, 3) | 1.682 (3.482) | 4.533 (4.536)
  Day 14 (n=10, 2) | -0.850 (1.255) | -0.650 (0.071)
  Day 21 (n=8, 2) | -0.825 (1.302) | -0.650 (0.071)
  Day 28 (n=9, 2) | 0.689 (1.279) | -0.650 (0.071)

28. Secondary Outcome: Numerical Pain Rating Scale (NPRS): Worst Pain (Weekly Average) in the Double-blind Treatment Period - AUC
Description: Participants assessed their pain levels by using the 0-10 Numeric Rating Scale: 0 = No pain 1-3 = Mild pain (nagging, annoying, interfering little with activities of daily living [ADLs]) 4-6 = Moderate pain (interferes significantly with ADLs) 7-10 = Severe pain (disabling; unable to perform ADLs A negative mean change denotes a pain decrease. A positive mean change denotes an increase in pain. Baseline was defined as the average of all measures taken from screening through the period prior to start of dosing on Day 1. Area under the curve (AUC) was computed using change from baseline in weekly average values at Day 7, Day 14, Day 21. and Day 28.
Time Frame: as for outcome 27
Measure: Mean (Standard Deviation); unit: NPRS score*week
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
NPRS score*week | -2.352 (2.674) | -3.229 (2.847)

29. Secondary Outcome: Numerical Pain Rating Scale (NPRS): Worst Pain (Weekly Average) in the Post-treatment Observation Period - Change From Baseline
Description: as for outcome 27
Time Frame: Participants assessed and recorded their pain level daily. Weekly averages were calculated for the Day 35, Day 42 and Day 49 assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post-treatment With Study Product Observation Period | Post-treatment With Placebo Observation Period
Number analyzed (Participants) | 10 | 2
score on a scale
  Day 35 (n=8, 2) | -4.675 (3.729) | -7.750 (1.202)
  Day 42 (n=10, 2) | -2.830 (5.494) | -7.750 (1.202)
  Day 49 (n=9, 2) | -3.089 (6.049) | -8.15 (0.212)

30. Secondary Outcome: Numerical Pain Rating Scale (NPRS): Worst Pain (Weekly Average) in the Post-treatment Observation Period - AUC
Description: Participants assessed their pain levels by using the 0-10 Numeric Rating Scale: 0 = No pain 1-3 = Mild pain (nagging, annoying, interfering little with activities of daily living [ADLs]) 4-6 = Moderate pain (interferes significantly with ADLs) 7-10 = Severe pain (disabling; unable to perform ADLs A negative mean change denotes a pain decrease. A positive mean change denotes an increase in pain. Baseline was defined as the average of all measures taken from screening through the period prior to start of dosing on Day 1. Area under the curve (AUC) was computed using change from baseline in weekly average values at Day 7, Day 14, Day 21, Day 28, Day 35, Day 42 and Day 49.
Time Frame: as for outcome 29
Measure: Mean (Standard Deviation); unit: NPRS score*week
Arm/Group | Post-treatment With Study Product Observation Period | Post-treatment With Placebo Observation Period
Number analyzed (Participants) | 10 | 2
NPRS score*week | -2.836 (3.637) | -6.118 (0.874)

31. Secondary Outcome: Numerical Pain Rating Scale (NPRS): Worst Pain (Weekly Average) in the Post-treatment Observation Period - Change From Last Day of Double-blind Treatment Period (Day 28)
Description: Participants assessed their pain levels by using the 0-10 Numeric Rating Scale: 0 = No pain 1-3 = Mild pain (nagging, annoying, interfering little with activities of daily living [ADLs]) 4-6 = Moderate pain (interferes significantly with ADLs) 7-10 = Severe pain (disabling; unable to perform ADLs A negative mean change denotes a pain decrease. A positive mean change denotes an increase in pain. Baseline was defined as the most recent value obtained on the last day of the double-blind dosing period (Day 28). Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: as for outcome 29
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post-treatment With Study Product Observation Period | Post-treatment With Placebo Observation Period
Number analyzed (Participants) | 10 | 2
score on a scale
  Day 35 (n=8, 2) | -3.425 (3.302) | -7.750 (1.202)
  Day 42 (n=10, 2) | -1.830 (4.905) | -7.750 (1.202)
  Day 49 (n=9, 2) | -1.978 (5.479) | -8.150 (0.212)

32. Secondary Outcome: Numerical Pain Rating Scale (NPRS): Worst Pain (Weekly Average) in the Post-treatment Observation Period - Change From Last Day of Double-blind Treatment Period (Day 28) - AUC
Description: Participants assessed their pain levels by using the 0-10 Numeric Rating Scale: 0 = No pain 1-3 = Mild pain (nagging, annoying, interfering little with activities of daily living [ADLs]) 4-6 = Moderate pain (interferes significantly with ADLs) 7-10 = Severe pain (disabling; unable to perform ADLs A negative mean change denotes a pain decrease. A positive mean change denotes an increase in pain. Baseline was defined as the most recent value obtained on the last day of the double-blind dosing period (Day 28). Area under the curve (AUC) was computed using change from baseline (Day 28) in weekly average values at Day 35, Day 42 and Day 49.
Time Frame: as for outcome 29
Measure: Mean (Standard Deviation); unit: NPRS score*week
Arm/Group | Post-treatment With Study Product Observation Period | Post-treatment With Placebo Observation Period
Number analyzed (Participants) | 10 | 2
NPRS score*week | -2.836 (3.637) | -6.118 (0.874)

33. Secondary Outcome: Brief Pain Inventory (BPI): Average Pain Level in Last 24 Hours (Double-blind Treatment Period) - Change From Baseline
Description: Participants rated the severity of their pain by using the BPI short form. Pain was rated on a scale from 0 (no pain) to 10 (pain as bad as you can imagine). A negative mean change denotes a pain decrease. A positive mean change denotes an increase in pain. Baseline was defined as the most recent value obtained prior to the start of the dosing on Day 1 of the double-blind dosing period. Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: At baseline, Day 7 and Day 28 during the double-blind treatment period
Population: Participants who provided baseline data and at least one other data point for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
score on a scale
  Day 7 (n=10, 3) | -0.4 (2.3) | -3.0 (3.3)
  Day 28 (n=8, 2) | -0.6 (1.2) | -1.3 (3.2)

34. Secondary Outcome: Brief Pain Inventory (BPI): Worst Pain Level in Last 24 Hours (Double-blind Treatment Period) - Change From Baseline
Description: as for outcome 33
Time Frame: At baseline, Day 7 and Day 28 during the double-blind treatment period
Population: Participants who provided baseline data and at least one other data point for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
score on a scale
  Day 7 (n=10, 3) | -1 (3) | 0 (0)
  Day 28 (n=8, 2) | -1 (3) | 1 (1)

35. Secondary Outcome: Brief Pain Inventory (BPI): Worst Pain Level in Last 24 Hours (Post-treatment Observation Period) - Change From Baseline
Description: Participants rated the severity of their pain by using the BPI short form. Pain was rated on a scale from 0 (no pain) to 10 (pain as bad as you can imagine). A negative mean change denotes a pain decrease. A positive mean change denotes an increase in pain. Baseline was defined as the most recent value obtained prior to the start of the dosing on Day 1 of the double-blind dosing period.
Time Frame: At baseline and Day 49 during the post-treatment observation period
Population: Participants who provided baseline data and at least one other data point for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post-treatment With Study Product Observation Period | Post-treatment With Placebo Observation Period
Number analyzed (Participants) | 8 | 2
score on a scale | -1 (5) | 0 (0)

36. Secondary Outcome: Brief Pain Inventory (BPI): Interference of Pain With Aspects of Life (General Activity) During Double-blind Treatment Period - Change From Baseline
Description: Participants rated the degree to which their pain interfered with various daily functions by using the BPI short form. Interference with general activity was rated on a scale from 0 (does not interfere) to 10 (completely interferes). Baseline was defined as the most recent value obtained prior to the start of the dosing on Day 1 of the double-blind dosing period. Category title includes number of participants with available data (n) for participants treated with study product, followed by participants treated with placebo.
Time Frame: At baseline, Day 7 and Day 28 during the double-blind treatment period
Population: Participants who provided baseline data and at least one other data point for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment With Study Product | Treatment With Placebo
Number analyzed (Participants) | 11 | 3
score on a scale
  Day 7 (n=10, 3) | 0 (2) | 0 (0)
  Day 28 (n=8, 2) | 1 (2) | 0 (0)

37. Secondary Outcome: Brief Pain Inventory (BPI): Interference of Pain With Aspects of Life (General Activity) During Post-treatment Observation Period - Change From Baseline
Description: Participants rated the degree to which their pain interfered with various daily functions by using the BPI short form. Interference with general activity was rated on a scale from 0 (does not interfere) to 10 (completely interferes). Baseline was defined as the most recent value obtained prior to the start of the dosing on Day 1 of the double-blind dosing period.
Time Frame: At baseline and Day 49 during the post-treatment observation period
Population: Participants who provided baseline data and at least one other data point for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Post-treatment With Study Product Observation Period | Post-treatment With Placebo Observation Period
Number analyzed (Participants) | 8 | 2
score on a scale | 0 (1) | 0 (0)

38. Secondary Outcome: Analgesic Use
Description: Analgesic use assessed with pain levels by numerical pain rating scale (NPRS) and brief pain inventory (BPI).
Time Frame: Throughout the study period (approximately 9 weeks)
Population: Data not collected for this outcome measure. Study terminated early.
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 0

39. Secondary Outcome: Reduction in Sickle Cell-specific Complications
Time Frame: Throughout the study period (approximately 9 weeks)
Population: Data not collected for this outcome measure. Study terminated early.
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Throughout study period (approximately 9 weeks)
Description: Summary tables for Adverse Events were provided per study period i.e. Placebo Lead-in Period, Double-blind treatment period and Post-treatment observation period. No breakdown of AEs with study product and placebo were provided as study terminated early.
Groups:
- Double-blind Treatment Period: Participants randomized 3:1 (Aes-103 to placebo) to receive 4 times daily dosing of either 1,000 mg of Aes-103 (study product) or placebo for 28 days (Day 1 to Day 28)
Arm/Group | Placebo lead-in Period | Double-blind Treatment Period | Post-treatment Observation Period
Serious Adverse Events (participants affected / at risk) | 2/23 | 0/14 | 1/12
Other Adverse Events (participants affected / at risk) | 21/23 | 12/14 | 4/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo lead-in Period (N=23) | Double-blind Treatment Period (N=14) | Post-treatment Observation Period (N=12)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 2 (2) | 0 (0) | 0 (0)
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo lead-in Period (N=23) | Double-blind Treatment Period (N=14) | Post-treatment Observation Period (N=12)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 13 (13) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (7) | 6 (6) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sickle cell anaemia (Congenital, familial and genetic disorders) | 5 (5) | 5 (6) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
PK data not determined as the assay collection method was found to be faulty rendering all samples unevaluable. Study was terminated early by the Sponsor due to unblinding between study drug and placebo groups at the subject, site and Sponsor levels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxalta's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, results may not be published without prior written approval of Sponsor.